CLINICAL TRIAL: NCT04385823
Title: Use of High Flow Nasal Cannula Oxygen During Acute Hypoxemic Respiratory Failure Related to Covid-19 and Interest of the Respiratory-oxygenation Index (ROX Index): an Observational Study
Brief Title: Use of High Flow Nasal Cannula Oxygen and Covid-19 Acute Hypoxemic Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Hôpital Louis Mourier (Other)
Responsible Party: Principal Investigator, Prof Jean-Damien RICARD, Head Medico-surgical ICU, Hôpital Louis Mourier
Other Study IDs: HLM_JDR9
Record Dates: First submitted 2020-05-11; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Syndrome, Acute, Severe; Hypoxic Respiratory Failure; Viral Pneumonia
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: patients receiving nasal high flow — patients admitted to the ICU for Covid-19-related acute hypoxemic respiratory failure treated with nasal high flow

SUMMARY:
Nasal High Flow oxygen therapy (NHF) is commonly used as first line ventilatory support in patients with acute hypoxemic respiratory failure (AHRF). It's use has been initially limited in Covid-19 patients presenting with AHRF. The aim of the study is to describe the use of NHF in Covid-19-related AHRF and report the changes in the respiratory-oxygenation index (termed ROX index) over time in these patients.

DETAILED DESCRIPTION:
Nasal High Flow oxygen therapy (NHF) is one of the newer methods of oxygenation commonly used in critical care during acute hypoxemic respiratory failure (AHRF). For various reasons (fear of a putative risk of viral dispersion; initial recommendations for rapid intubation due to the rapid deterioration of patients), NHF seems to have been seldomly used during the current Covid-19 epidemic in France. However, the World Health Organization, and other scientific societies list NHF among the possible options for ventilatory support.

One of the risks however, identified with NHF is to delay an intubation that would have become necessary. This delay seems to be associated with a poorer prognosis for patients.

The respiratory-oxygenation index (termed ROX index) (defined as the ratio of pulse oximetry (SpO2) over inspired fraction in oxygen (FiO2) over respiratory rate (RR); SpO2/FiO2/RR) is used - along with other criteria - to assist the clinician in deciding whether or not to intubate patients on NHF for AHRF. In investigators'ICU, NHF is used in patients admitted for AHRFrelated to Covid-19 and the ROX index is measured and monitoring in investigators' patients. Investigators' initial experience - consistent with feedback from other ICUs - suggests that the respiratory rate of patients with Covid-19-related AHRF is sometimes lower than would be expected given the depth of the hypoxemia. In this case, the ROX index thresholds previously identified for predicting the success or failure of NHF could be different in the case of Covid-19-associated AHRF. The purpose of this work is to describe the use of NHF in Covid-19 patients with AHRF and the evolution of the ROX score over time in patients initially treated with NHF.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 pneumonia
* acute hypoxemic respiratory failure
* need for nasal high flow therapy as first line therapy
* admission to intensive care

Exclusion Criteria:

* intubation prior to NHF therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients admitted to the ICU with proven Covid-19 pneumonia and acute hypoxemic respiratory failure requiring supplemental oxygen administered via NHF
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Changes in ROX index | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  values of ROX index during ICU stay

SECONDARY OUTCOMES:
NHF failure | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  percentage of patients requiring intubation
NHF flow | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  level of flow used with NHF
NHF inspired fraction in oxygen | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  level of inspired fraction in oxygen used with NHF
oxygenation | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  level of pulse oxymetry during NHF therapy
respiratory status | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  respiratory rate during NHF therapy
prediction of intubation | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  defining the values of ROX index associated with intubation
prediction of NHF success | from date of NHF initiation until date of weaning from NHF or date of intubation whichever came first, assessed up to 2 months
  defining the values of ROX index associated with NHF success (no intubation required)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Damien Ricard, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Louis Mourier, Assistance Publique - Hôpitaux de Paris, Colombes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760